Official Title: Effect of supplementation with *Euterpe edulis* on the physical and mental performance of healthy men subjecting to physical exercise

Ethical committee Protocol No: 6.202.888

Inform consent



Document date: September 15th, 2023

## **INFORM CONSENT TERM (TCLE)**

Effect of supplementation with *Euterpe edulis* on the physical and mental performance of healthy men subjecting to physical exercise Responsible for research: Prof. Dr Denise Coutinho Endringer

This document you are reading is called the Free and Informed Consent Term (TCLE). It contains explanations about the study you are being asked to attend. Before deciding whether to participate (of your own free will) you should read and understand all the content. In the end, if you decide to participate, you will be asked to sign it and you will receive a copy of it. Before signing, ask questions about anything you did not understand well. The study team will respond to your questions at any time (before, during and after the study). Your participation is voluntary, which means that you can withdraw at any time, withdrawing your consent, without any loss or penalty, by contacting one of the responsible researchers.

This research seeks to evaluate the capacity for muscle recovery with the use of juçara juice. If you decide to accept the invitation, you will drink a dose of juçara juice daily for a period of 10 days and biochemical tests will be collected before and after performing the physical exercise. In addition, the participant will answer questionnaires before and after consuming the juice to assess intestinal functioning and microbiota. It is expected that the consumption of juçara juice will be able to reduce the time of fatigue, pain and exhaustion after physical exercise.

The risks that may occur when carrying out such research are related to the leakage of the individual's private information and this data being used by third parties, which is avoided by using passwords to access the data. If this procedure can generate some kind of embarrassment, you do not have to do it.

You will have the following benefits by participating in this research: Studies indicate that a diet enriched with juçara juice can preserve spontaneous motor performance, increase exploration in the aversive environment (anxiolytic-like

effects) and increase the latency to step-down (better retention memory), in addition to reducing the level of lipid peroxidation in the hippocampus. If this data is proven, you may benefit in these aspects.

All information obtained will be confidential. The material with your information will be kept in a safe place under the responsibility of the main researcher represented by Dr. Denise Coutinho Endringer, with the guarantee of maintaining secrecy and confidentiality and will be destroyed after the research. The results will be published in a way that does not identify the volunteers. The results of this work may be presented at meetings or scientific journals, however, it will only show the results obtained as a whole, without revealing its name, the institution to wich it belongs or any information related to its privacy.

As provided by the Brazilian research standards with the participation of human beings you will not receive any type of financial compensation for your participation in this study. If you have any expense that is due to your participation in the survey, you will be reimbursed if you request it. At any time, if you experience any damage from this research, you will be entitled to compensation.

You will be left with a route to this Term and any questions you have regarding this research, you can ask directly to the researcher Deuel Azolin Da Silva: (27) 98166-9697 or to the Rectory Building Committee – Underground Avenida Comissário José Dantas de Melo, n°21, Boa Vista, Vila Velha-ES, CEP: 29.102-920, Tel: (27) 3421-2063 E-mail: CEP@uvv.br

Opening hours: Monday to Thursday 7am to 12pm and 1pm to 5pm and Friday - 7am to 12pm and 1pm to 4pm. Complaints and/or dissatisfaction related to the patient's participation in the research may be communicated in writing to the CEP/UVV Secretariat, provided that the claimants identify themselves, and their name will be kept anonymous.

## Consent

| Signature of the Principal Investigator: | Date |
|------------------------------------------|------|
| Signature of the Patient: | Date |